CLINICAL TRIAL: NCT05243667
Title: Research on the Early Warning Model of Children Asthma Acute Attack Based on Wearable Wrist Smart Device of Huami
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, LI-HONG SUN, Clinical Professor, Guangzhou Institute of Respiratory Disease
Other Study IDs: GuangzhouIRD-LSUN2
Record Dates: First submitted 2021-08-15; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Asthma in Children
Keywords: Wearable wrist Smart Device

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Wearable wrist Smart Device of Huami — All enrolled patients underwent continuous monitoring by wearing huami blood oxygen testing equipment, and signed the informed consent for the clinical trial.Smart wrist wristbands will be issued, and patient information will be bound to the "Migang Health" platform, and clinical trial doctors will improve relevant personal information and clinical data.After binding to the APP "Migu Health", you can start collecting and recording dynamic data such as peripheral blood oxygen saturation, heart rate, exercise steps, sleep data, etc., and upload the data once a day.

SUMMARY:
Childhood asthma is the most common chronic respiratory disease in childhood. The essence of asthma is chronic airway inflammation and airway hyperresponsiveness.The physiological characteristics of children and adults are very different, and the compensatory ability is very strong. There are often no obvious symptoms at the early stage of attack, or only intermittent or persistent cough of different degrees, without typical chest tightness and asthma.However, at this time, certain physiological indicators such as blood oxygen, heart rate, respiratory rate may have been significantly abnormal.If the disease continues to deteriorate and progresses to decompensation, it can quickly move from an asymptomatic state to a failure stage.Therefore, dynamic and accurate acquisition of real-time vital signs and assessment is of great significance for early warning and improvement of prognosis of asthma attacks in children.Intelligent wearable devices can be used to acquire real-time physiological index data of users, such as heart rate, blood oxygen, exercise and sleep dynamic data.An in-depth analysis of long-term and multi-scene dynamic data before and after asthma attacks can establish an early warning model for children with acute asthma attacks by wearable wrist smart devices, which may provide important help for severity assessment, follow-up tracking and out-of-hospital prevention and control of the disease.

DETAILED DESCRIPTION:
this project is selected 200 cases of children with asthma diagnosis definitely, collection and heart rate, blood oxygen, exercise and sleep dynamic data, followed up for 3 to 6 months (at least 3 months), records of clinical asthma attacks and clinical data, through the cloud data analysis and deep learning, analysis of children with asthma attacks and multiple physiological parameters (heart rate, blood oxygen, movement and the dynamic data of sleep, etc.), the connection between the building of asthma early warning and illness severity hierarchical evaluation model.Then choose 200 cases of diagnosis in clinical practice to determine follow-up, patients with asthma children to observe to verify the exactness of the model of asthma attack early warning, and according to the collected data to further improve, calibration model, designed to provide children with family members and medical personnel of an asthma attack warning and follow-up management wearable auxiliary equipment and management platform.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of asthma.

Exclusion Criteria:

Severe chronic diseases with organ dysfunction and dyspnea.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with diagnosed asthma.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Heart rate | up to 24 weeks
  Follow-up monitoring of confirmed asthma patients was conducted based on intelligent wearable devices, and multiple physiological parameters such as heart rate were collected in the pre-attack, attack and remission stages
blood oxygen | up to 24 weeks
  Follow-up monitoring of confirmed asthma patients was conducted based on intelligent wearable devices, and blood oxygen were collected in the pre-attack, attack and remission stages
exercise | up to 24 weeks
  Follow-up monitoring of confirmed asthma patients was conducted based on intelligent wearable devices, and exercise were collected in the pre-attack, attack and remission stages
sleep | up to 24 weeks
  Follow-up monitoring of confirmed asthma patients was conducted based on intelligent wearable devices, and sleep were collected in the pre-attack, attack and remission stages

SECONDARY OUTCOMES:
weight | up to 24 weeks
  Weight of enrolled asthmatic patients
height | up to 24 weeks
  Height of enrolled asthmatic patients

CONTACTS AND LOCATIONS:
Overall Officials: Qin C Pan, master, Principal Investigator — Guangzhou Institute of Respiratory Disease
Locations (1):
- Guangzhou institute of respiratory disease, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Within six months after the trial complete.

REFERENCES:
- [Result] Kumar N, Akangire G, Sullivan B, Fairchild K, Sampath V. Continuous vital sign analysis for predicting and preventing neonatal diseases in the twenty-first century: big data to the forefront. Pediatr Res. 2020 Jan;87(2):210-220. doi: 10.1038/s41390-019-0527-0. Epub 2019 Aug 4. PMID 31377752
- [Result] Jensen CS, Aagaard H, Olesen HV, Kirkegaard H. A multicentre, randomised intervention study of the Paediatric Early Warning Score: study protocol for a randomised controlled trial. Trials. 2017 Jun 8;18(1):267. doi: 10.1186/s13063-017-2011-7. PMID 28595614
- [Result] Carew C, Cox DW. Laps or lengths? The effects of different exercise programs on asthma control in children. J Asthma. 2018 Aug;55(8):877-881. doi: 10.1080/02770903.2017.1373806. Epub 2017 Oct 16. PMID 28872938